CLINICAL TRIAL: NCT04703374
Title: A Randomized, Open-label, Crossover Phase 1 Clinical Trial to Compare Pharmaciokinetics, Pharmacodynamics and Safetry After Single/ Multiple Administration of CKD-382 and D026 in Healthy Subjects
Brief Title: A Study to Compare PK, PD and Safety of CKD-382 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A105_01BE2010
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: GERD
Keywords: CKD-382; D026
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- A (Experimental): Period 1: Test drug(CKD-382 formulation I) Period 2: Test drug(CKD-382 formulation II) Period 3: Reference drug(D026)
  Interventions: Drug: CKD-382(formulation I); Drug: CKD-382(formulation II); Drug: D026
- B (Experimental): Period 1: Test drug(CKD-382 formulation II) Period 2: Reference drug(D026) Period 3: Test drug(CKD-382 formulation I)
  Interventions: Drug: CKD-382(formulation I); Drug: CKD-382(formulation II); Drug: D026
- C (Experimental): Period 1: Reference drug(D026) Period 2: Test drug(CKD-382 formulation I) Period 3: Test drug(CKD-382 formulation II)
  Interventions: Drug: CKD-382(formulation I); Drug: CKD-382(formulation II); Drug: D026
- D (Experimental): Period 1: Test drug(CKD-382 formulation I) Period 2: Reference drug(D026) Period 3: Test drug(CKD-382 formulation II)
  Interventions: Drug: CKD-382(formulation I); Drug: CKD-382(formulation II); Drug: D026
- E (Experimental): Period 1: Test drug(CKD-382 formulation II) Period 2: Test drug(CKD-382 formulation I) Period 3: Reference drug(D026)
  Interventions: Drug: CKD-382(formulation I); Drug: CKD-382(formulation II); Drug: D026
- F (Experimental): Period 1: Reference drug(D026) Period 2: Test drug(CKD-382 formulation II) Period 3: Test drug(CKD-382 formulation I)
  Interventions: Drug: CKD-382(formulation I); Drug: CKD-382(formulation II); Drug: D026

INTERVENTIONS:
Drug: CKD-382(formulation I) — 1 tablet administered under fasting condition for 7days
Drug: CKD-382(formulation II) — 1 tablet administered under fasting condition for 7days
Drug: D026 — 1 tablet administered under fasting condition for 7days

SUMMARY:
To compare pharmacokinetics, pharmacodynamics and safety after single/multiple administration of CKD-382 and D026 in healthy subjects

DETAILED DESCRIPTION:
A randomized, open-label, crossover phase 1 clinical trial to compare pharmacokinetics, pharmacodynamics and safety after single / multiple administration of CKD-382 and D026 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

1. Between 19 aged and 50 aged in healthy adult
2. Body weight more than 50kg
3. Body Mass Index more than 18.0 and under 27.0
4. Who has negative result on Helicobacter Pylori antibody test

Exclusion Criteria:

1. Have clinically significant disease that hepatobiliary system, kidney, nervous system, immune system, respiratory system, endocrine system, hemato-oncology disease, cardiovascular system or mental illness, or a history of mental disease.
2. Have a gastrointestinal disease history(including surgery) that can effect drug absorption
3. Hypersensitivity reaction or clinically significant hypersensitivity reaction in the history of Esomeprazole, additives or benzimidazole family.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-09-25 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
AUCtau,ss(Area under the plasma drug concentration-time curve within a dosing interval at steady state) Evaluation PK after multiple dose | 0~24h
Percent decrease from baseline in integrated gastric acidity for 24-hour interval after 7th dose Evaluation PD for ambulatory 24hr pH monitor | Baseline versus Multiple dose during 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Chungbuk National University Hospital, Cheongju-si, North Chungcheong, South Korea

IPD SHARING:
Plan to Share IPD: No